CLINICAL TRIAL: NCT04901819
Title: Longterm Outcomes of Individuals With Anorectal Malformations
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Tomas Wester, Professor, Karolinska Institutet
Other Study IDs: FOR 4-1500/2021; K 2021-4578 (Other: Karolinska University Hospital)
Record Dates: First submitted 2021-05-19; First posted 2021-05-26 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Anorectal Malformations
MeSH Terms: conditions — Anorectal Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a cross-sectional observational study with the aim to assess longterm outcomes in a large cohort of individuals with anorectal malformations. Patients managed for anorectal malformations at Karolinska University Hospital, Stockholm, Sweden, Stockholm 1994-2017 will be reviewed and they will be invited to respond to validated questionnaires evaluating bowel function (>4 years of age), urinary tract function (>4 years of age), sexual function (>18 years of age) and quality of life (>8 years of age). Data will be analyzed with descriptive and comparative statistics.

DETAILED DESCRIPTION:
Background Anorectal malformations comprise a spectrum of congenital anomalies, that range from mild anterior displacement of the anus to very complex anomalies, involving both the hindgut and the urogenital tract. The birth prevalence in Sweden is approximately 1:3000 (1). Associated anomalies are encountered in 50-60 % of individuals with anorectal malformation. Anorectal malformations are associated with tethered cord in 20-30% of patients, which may impair bowel and urinary tract function. Development of surgical techniques and neonatal care have improved survival of children with anorectal malformations over the last decades. The focus of care has shifted from survival to optimizing bowel and urinary tract function as well as reducing the negative impact on quality of life. Current surgical techniques were introduced during the early 1980's. The outcomes compare favorably with older techniques, although there is still limited information on the outcomes up to adult age. Particularly, there are limited data of composite outcomes of bowel function, urinary tract function, sexual function and quality of life in comparison to age- and gender-matched controls from the normal population. Newborn infants are often screened for tethered cord with ultrasound. It is unclear if infants with normal ultrasound also need an MRI at a later stage to exclude spinal cord anomalies. Tethered cord is frequently asymptomatic. There are conflicting data with respect to prophylactic de-tethering.

Aims The overall aim of this project was to assess composite outcomes, bowel function, urinary tract function, sexual function, and quality of life in a cross-sectional study of children with ARM managed at Karolinska University Hospital.

Specific aims

1. To assess if bowel function, urinary tract function, sexual function, and quality of life is impaired in children with ARM compared with normative data.
2. To assess if bowel function, urinary tract function, sexual function and quality of life correlate
3. To assess if individuals with ARM and tethered cord benefit from detethering.
4. To assess if ultrasound of the spinal cord and MRI are equal imaging modalities to diagnose tethered cord.

Methods Study design Cross-sectional observational study. The STROBE Statement for reporting of observational studies will be used (2).

Settings and participants All individuals managed for an anorectal malformation at Karolinska University Hospital from 1994 to 2017 will be eligible for the study. Patients and/or parents who provide informed consent and fill in the questionnaires will be included in the study. There will be 300-400 eligible patients.

Data sources and variables Demographic and clinical details will be recorded retrospectively from the medical records, including gender, birth weight, gestational age, associated syndromes and anomalies, family history, presenting symptoms, type of ARM, surgical details including postoperative complications and re-operations. Questionnaires will be sent according to age to the participants to assess bowel function, urinary tract function, sexual function, and quality of life. Questionnaires on sexual function and quality of life will not be sent to individuals with intellectual impairment, eg. Down syndrome. It will be possible to respond to the questionnaires using a digital platform. Bowel function will be assessed in individuals more than 4 years of age using a bowel function score (BFS) questionnaire (3) developed for assessment of bowel function in pediatric anorectal disorders and validated in patients and in the general Finnish population (4). Urinary tract function will be assessed in individuals more than 4 years of age with a questionnaire on lower urinary tract symptoms, with questions addressing history of urinary tract infection, urgency, urge incontinence, stress incontinence, straining to begin urination, and leakage of urine without physical activity or apparent need to urinate, based on items adapted from the previously validated Danish Prostatic Symptom Score. Profile of Sexual Female function will be used to assess sexual function in the female patients more than 18 years of age. IIEF will be used to assess sexual function in males more than 18 years of age. KIDSCREEN, a validated instrument assessing children's and adolescents subjective health and well-being, will be used to assess the quality of life in children and adolescents 8 to 18 years of age. In patients more than 18 years old, Psychological general well-being index (PGWB) will be used to assess quality of life. In a sub-study, individuals with tethered cord will be identified. The outcomes among patients with tethered cord who have undergone de-tethering will be compared with those who have not undergone an operation. In a second sub-study, spinal cord ultrasound and MRI images will be reviewed by two experienced pediatric radiologists in a blinded fashion. Correlation between the two imaging modalities will be analyzed.

Data analysis Pseudonymized data will be recorded in Excel spread sheets. Data will be analyzed with descriptive and comparative statistics. Matched controls and normative population-based data will be used for comparison.

Ethics Patients and/or caregivers will receive written information about the study and provide written informed consent. Data that are entered into the project database will be pseudonymized to protect privacy. The benefit of the study are considered to exceed the risks.

Significance The knowledge of long-term outcomes up to adulthood in patients with anorectal malformations is limited. Particularly controlled data are scanty. This study may contribute important additional understanding and contribute to improved care of individuals with anorectal malformations.

Project timeline Autumn 2020: Ethical approval application. Identification of eligible patients. Spring 2021: All patients will be invited to participate and questionnaires sent out. Data collection.

Autumn 2021- 31 December 2026: Data collection. Collected data will be analysed and summarized in publications.

ELIGIBILITY:
Inclusion Criteria:

Individual who has undergone surgical management for anorectal malformation at Karolinska University Hospital 1994 to 2017.

Exclusion Criteria:

Individual not providing informed consent.

Ages: 4 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individual who have undergone surgical management for anorectal malformations at Karolinska University Hospital, Stockholm, Sweden from 1994 to 2017.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Bowel function score | 3 years
  Bowel function score, BFS, >4 years of age (Rintala et al. J Pediatr Surg 1995;30:491-4)
Urinary tract function | 3 years
  Urinary tract function evaluated with a modification of Danish Prostatic Symptom Score, >4 years of age (Kyrklund et al Dis Colon Rectum 2012;55:671-6)
Sexual function | 3 years
  Sexual function evaluated with Profile of Female Sexual Function in females >18 years of age and with IIEF in males >18 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Wester, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Svenningsson A, Gunnarsdottir A, Wester T. Maternal risk factors and perinatal characteristics of anorectal malformations. J Pediatr Surg. 2018 Nov;53(11):2183-2188. doi: 10.1016/j.jpedsurg.2018.04.021. Epub 2018 Apr 17. PMID 29907315
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739
- [Background] Rintala RJ, Lindahl H. Is normal bowel function possible after repair of intermediate and high anorectal malformations? J Pediatr Surg. 1995 Mar;30(3):491-4. doi: 10.1016/0022-3468(95)90064-0. PMID 7760250
- [Background] Kyrklund K, Koivusalo A, Rintala RJ, Pakarinen MP. Evaluation of bowel function and fecal continence in 594 Finnish individuals aged 4 to 26 years. Dis Colon Rectum. 2012 Jun;55(6):671-6. doi: 10.1097/DCR.0b013e31824c77e4. PMID 22595847